CLINICAL TRIAL: NCT03023670
Title: Ventilatory Patterns During Cardiopulmonary Bypass In Pediatric Cardiac Surgery
Brief Title: Lung Protection and Pediatric Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sayed Kaoud Abd-Elshafy, Associate profossor of anesthesiology and critical care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB0000871180
Record Dates: First submitted 2017-01-11; First posted 2017-01-18 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Lung Injury, Acute
Keywords: Lung; Cardiopulmonary Bypass; Pediatric; Cardiac surgery
MeSH Terms: conditions — Acute Lung Injury | interventions — Cardiopulmonary Bypass; Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): This group will include patients with low flow of mixed oxygen / air (1:1L) during the period of cardiopulmonary bypass
  Interventions: Procedure: cardiopulmonary bypass
- Group B (Active Comparator): This group will receive low rate (4\min) with low tidal volume ( 2ml/kg ) during the period of cardiopulmonary bypass.
  Interventions: Procedure: cardiopulmonary bypass

INTERVENTIONS:
Procedure: cardiopulmonary bypass — Low flow of mixed oxygen / air (1:1L) will be used during the period of cardiopulmonary bypass
  Other Names: Control group
  Arms: Group A
Procedure: cardiopulmonary bypass — Low rate (4\min) with low tidal volume ( 2ml/kg ) will be used during the period of cardiopulmonary bypass.
  Other Names: Low frequency group
  Arms: Group B

SUMMARY:
The lung is at risk for ischemic insults during total cardiopulmonary bypass because lung perfusion is maintained solely by the bronchial arterial system

DETAILED DESCRIPTION:
The study will be performed in the pediatric cardiothoracic unit, pediatric Assiut University Hospital. After obtaining approval from the local ethics committee and written informed parents consent 60 patients will be included in this study according to the following criteria:

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgery
* Ventricular septal defect (VSD).
* Atrial septal defect (ASD)

Exclusion Criteria:

* Cyanotic heart disease.
* Patients with preoperative chest problems.
* Patients with known renal or hepatic dysfunctions.
* Planned off-pump cardiac surgery.
* Emergency cardiac surgery.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Computerized tomography chest (CT chest) within 7 days postoperative | preoperative and within the first 7 days postoperative

SECONDARY OUTCOMES:
Mechanical ventilation | Within the first 7 days postoperative
  Duration of mechanical ventilation (hours)
Intensive care unit stay | Within the first 7 days postoperative
  Intensive care unit stay
Intubation time | Within the first 7 days postoperative
  Intubation time (hours)
Arterial blood gases | Within the first 7 days postoperative
  Intraoperative and postoperative by appropriate scale

CONTACTS AND LOCATIONS:
Overall Officials: Sayed Abd-Elshafy, M.D, Principal Investigator — Associate profossor of Anesthesiology and critical care
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided